CLINICAL TRIAL: NCT05240495
Title: Work-focused Versus Generic Internet-based Interventions for Employees With Stress-related Disorders - a Randomized Controlled Trial
Brief Title: Work-focused Versus Generic Internet-based Interventions for Stress-related Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Gerhard Andersson, Professor, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: iStress3
Record Dates: First submitted 2022-01-15; First posted 2022-02-15 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Adjustment Disorders
Keywords: Stress; Burnout; Exhaustion; Work-focused; Internet-based; Sickness absence
MeSH Terms: conditions — Adjustment Disorders; Burnout, Psychological

STUDY DESIGN:
Intervention Model Description: This study was a three-armed controlled superiority trial in which two internet-based interventions for stress-related disorder: (a) cognitive-behavioural therapy (iCBT; n=61) and (b) work-focused iCBT (W-iCBT; n=61) that integrated work aspects early into the treatment, were compared against a wait-list control group (n=60). The study followed the CONSORT guidelines [45]. Sample size was estimated on the basis of previous controlled trials on iCBT for chronic stress (e.g., Persson Asplund et al., 2018), with the aim of detecting an effect size of Cohens'd=0.50 on the primary outcome Shirom-Melamed Burnout Questionnaire (see Measures), at post assessment, based on a power of 0.80 in a two-tailed test with 0.05 significant level. Self-reported outcome assessments were collected at pre- and post-treatment (ten weeks) and at a 6- and 12-month follow-up.
Who Masked: Participant
Masking Description: Single blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Internet-based Cognitive-behavioural therapy group (n=61) (Experimental): TThe generic iCBT program was based on contemporary CBT techniques adapted for stress-related disorders, and recovery from work training inspired by Hahn et al. [2011]. The iCBT consisted of ten modules distributed over ten weeks, with modules lasting 60-120 min per week. In the first module (introduction), the participants received information about the outline of the program, stress physiology and defined individual treatment goals. During the second week participants were introduced to different recovery techniques and applied relaxation. The third and fourth week contained exercises related to behavioral activation, work-home balance, and values-based action skills. Between weeks five and ten, participants were able to choose between different exposure-based exercises. In addition, participants with insomnia could choose to focus on sleep management.
  Interventions: Behavioral: Internet-based Cognitive-behavioural therapy
- Internet-based Work-focused Cognitive-behavioural therapy group (n=61) (Experimental): The internet-based and work-focused cognitive-behavioral therapy (W-iCBT) consisted of the generic treatment for stress-related disorders (iCBT), plus components focusing on work and return-to-work. These sections were integrated and represented in each of the ten modules. Work-focused CBT is built on the same conceptual framework as regular CBT. For example, CBT principles are used to change the appraisal of work stressors, change the dysfunctional behaviour, or increase health promoting behaviours. The CBT principal, exposure, is given special attention. Gradual exposure can help individuals develop more effective coping skills when dealing with work-related stressors (e.g., assertiveness) and stimulate gradual return to the work setting for individuals on a long-term sick leave [27].
  Interventions: Behavioral: Internet-based Cognitive-behavioural therapy; Behavioral: Work-focused Cognitive-behavioural therapy
- Wait-list control group (n=60) (No Intervention): Wait-list control group received equal and parallell assessment and eligibility procedure as the two experimental konditions. Wait-list control group gained access to iCBT/W-iCBT program after the six months follow-up.

INTERVENTIONS:
Behavioral: Internet-based Cognitive-behavioural therapy — Internet-based Cognitive-behavioural therapy protocol was based on contemporary CBT techniques adapted for adjustment disorders, and recovery from work training inspired by Hahn et al. [50]. The iCBT program consisted of ten modules distributed over ten weeks, with modules lasting 60-120 min per week.
  Arms: Internet-based Cognitive-behavioural therapy group (n=61); Internet-based Work-focused Cognitive-behavioural therapy group (n=61)
Behavioral: Work-focused Cognitive-behavioural therapy — The Work-focused Cognitive-behavioural therapy consisted of the exact generic iCBT-modules included in the first experimental group and of additional work-focused modules adapted for adjustment disorders. The W-iCBT added about 2-3 regular pages compared to the generic iCBT.
  Arms: Internet-based Work-focused Cognitive-behavioural therapy group (n=61)

SUMMARY:
Objective The aim of the current study was to evaluate the efficacy of an internet-based cognitive-behavioural intervention for stress-related disorders integrating work-related aspects (W-iCBT), compared with a generic iCBT and a waitlist control group (WLC).

Method In this trial, 182 employees, mainly employed in the healthcare, IT or educational sector, who fulfilled the criteria for a stress-related disorder, were randomized to a 10-week W-iCBT (n=61), generic iCBT (n=61) or WLC (n=60). Self-rated questionnaires on perceived stress, burnout, exhaustion and other mental-health and work-related outcomes were administered pre- and post-treatment, and at a six- and 12-months follow-up.

Results Compared to WLC, participants of the W-iCBT and iCBT showed equal and significant reduction on the primary outcome (SMBQ) from pre to post assessment (d=1.00 and 0.83 respectively) and at the six months follow-up (d=0.74 and 0.74). Significant moderate-to-large effect sizes were also found on the secondary health and work-related outcomes. The W-iCBT was the only group who exhibited significant effects on work ability and sickness absence. Sickness absence was 445 days (7.29 days per participant) lower compared to the WLC and 324 days (5.31 days per participant) compared to the iCBT intervention. However, no significant differences were found on work experience or long-term sick leave.

Conclusion The work-focused and generic iCBT interventions proved to be superior and equally effective compared to the control condition in reducing chronic stress and several other mental health related symptoms. Interestingly, effects on work ability and sickness absence were only seen between the work-focused iCBT intervention and the WLC. These preliminary results are promising, as they provide further evidence that treatments that integrate work-aspects has great potential in accelerating both recovery and reduce sickness absence due to stress-related disorders.

DETAILED DESCRIPTION:
Introduction Work is an important part of life, contributing to both health and wellbeing for many employees. However, in recent years, stress-related disorders have received more attention, with an increasing prevalence within the working population. For example, every fourth employee within the European union has experienced stress during most of their working day. Long-term exposure to stressors, such as job strain or interpersonal conflicts, without sufficient recovery, can lead to a dysregulation in the allostatic system, "allostatic load", which constitutes the fundamental features in the development of chronic stress or stress-related disorders. The major diagnostic systems, Diagnostic and Statistical Manual of Mental Disorders (DSM-5) and International Statistical Classification of Diseases and Related Health Problems (ICD-10 and 11) includes sections regarding stress-related disorders. However, the DSM and ICD systems lack an established terminology and criteria for stress induced fatigue and exhaustion. Consequently, the diagnosis "Exhaustion disorder" (ED) was introduced in the Swedish version of the ICD-10 in 2005. ED is manifested by symptoms of extensive mental and physical fatigue, lack of initiative and endurance and prolonged recovery after mental or physical effort. Later international publications have suggested that ED is not an exclusive Swedish condition. Few studies have been published regarding the prevalence of ED, but in a recent study, based on physician-based diagnosis in 3406 participants, 4.2% reported ED.

In addition to stress-related disorders and well-known health implications, such as coronary artery disease, lowered immune functioning, anxiety, depression and insomnia, chronic stress have been associated with impaired work functioning and problems in work participation such as sickness absence and long-term sick leave. In Sweden, for example, stress-related disorders accounted for one fifth of all sick leave during 2019. Decreased work participation is problematic as it has direct effects on people's well-being and leads to immense costs for society. For instance, the total estimated annual costs for work-related stress observed in seventeen OECD countries is considerable, ranging from US $221 million to $187 billion. Given these rising costs, it is not surprising that many policy makers view stress as a major public health issue and are seeking advice on the types of interventions that may be effective.

During the last decades, psychological interventions have been developed in order to increase the individual's psychological resources and resilience to stress. Evidence suggest that stress management interventions are effective in reducing stress in the working population. These results apply to controlled studies targeting general and milder forms of stress-related ill health. However, considering clinical samples, interventions has been less successful, with small effect sizes.

Traditionally, psychological treatments for stress and common mental disorders have not explicitly focused on work-related aspects, such as reducing sickness absence (SA). Recent evidence suggests that psychological interventions are slightly more effective than treatment-as-usual in reducing sickness absence (small effect sizes). However, it is still uncertain what moderates these effects. There are some indications that work directed interventions in combination with psychological treatment are effective with respect to return-to-work (RTW) for those absent with common mental health problems. In a quasi-experimental study by Lagervelt and colleagues comparing CBT to work-focused CBT, full RTW occurred 65 days earlier and partial RTW 12 days earlier in the work-focused CBT group. A significant decrease in mental health problems was equally present in both conditions. These results suggest that by integrating work-related aspects early into the treatment, problems with sickness absence and long-term sick leave can be reduced.

Despite the well-documented efficacy of stress management interventions, and some promising results of work-focused interventions, the range of interventions are not proportionate to the needs among distressed employees. This clarifies the need to further develop and evaluate work directed interventions that are accessible to the working population.

Studies suggest that stress can be managed through internet- and computer-based interventions. In a meta-analysis including 26 controlled studies (n=4226), small to moderate effects were found on outcomes on stress, depression and anxiety. Subgroup analyses revealed that guided interventions were more effective. Studies also suggest that internet-based interventions for stress can have sustained effects on stress reduction, be cost-effective, and have positive effects on participant's experiences on health and wellbeing in both work and private life. However, previous iCBT studies have focused on individuals with elevated stress and few studies has evaluated the efficacy of iCBT in clinical samples, such as employees with stress-related disorder. In addition, we found no previous studies evaluating the efficacy of internet-based and work-focused interventions on sickness absence and RTW.

Purpose of the present study The aim of the current study was to evaluate the efficacy of iCBT for stress-related disorders integrating work-related aspects (W-iCBT) and a generic iCBT, compared to a waitlist control condition (WLC). We hypothesized that W-iCBT and iCBT would be superior and equally effective in reducing perceived stress, burnout, exhaustion, and improving recovery from work and quality of life, compared to a WLC. In secondary explorative analyses, we examined whether the W-iCBT would differ from the iCBT and WLC with regard to important work-related outcomes including work experience, work ability, sickness absence and long-term-sick-leave. We also hypothesized that initially achieved changes would remain stable at a 12-month follow-up.

Method

Design This study was a three-armed controlled superiority trial in which two internet-based interventions for stress-related disorder: (a) cognitive-behavioural therapy (iCBT) and (b) work-focused iCBT (W-iCBT) that integrated work aspects early into the treatment, were compared against a wait-list control group. The study followed the CONSORT guidelines. Sample size was estimated on the basis of previous controlled trials on iCBT for chronic stress, with the aim of detecting an medium effect size on the primary outcome Shirom-Melamed Burnout Questionnaire (see Measures), at post assessment, based on a power of 0.80 in a two-tailed test with 0.05 significant level. Self-reported outcome assessments were collected at pre- and post-treatment (ten weeks) and at a 6- and 12-month follow-up. Participants who met the study criteria and provided informed consent were randomly allocated by an independent researcher using an internet-based random generator (www.randomizer.org). The independent researcher received a list of anonymous identification numbers of all participants and coaches. This procedure ensured that blinding was implemented during randomization. All participants, coaches and those participants reporting benefits due to long-term sick leave at baseline, were randomized in a 1:1:1 proportion. The Ethical Committee of Linkoping University, Sweden, approved all procedures involved in the study (reference number 2016/11-31).

Procedure The study was conducted in a university setting, with researchers and the treatment platform hosted by the university. Participants were recruited from the general public through advertisement, articles in regional and national newspapers, and labour organization magazines. Detailed information and application to the study was presented on the project's homepage (www.istress.se). After initial registration using personal e-mail address, potential participants received an ID number and were asked to (i) provide written informed consent, (ii) complete online screening questionnaires (see Measures) and (iii) participate in a diagnostic interview over the telephone. Following the interview, the included participants were randomized. Participants of the iCBT and W-iCBT groups received access to the programs immediately after randomization and participants of the wait-list control group received access to iCBT/W-iCBT program after the six months follow-up.

Support Every week, participants in both interventions (W-iCBT and iCBT) received personalized written messages from a coach with feedback on the exercises. For the participants in the W-iCBT group, guidance was given on the CBT and work-focused modules simultaneously. The coaches, eight in total, were master level psychology students who were specifically trained to perform feedback according to a standardized manual. The aim of the feedback was to provide support and encouragement and to monitor homework assignments and adherence to the intervention. Treatment as usual was not prohibited but also not encouraged during the trial. The coaches were requested to minimize their support to one message and 15 min of correspondence per week and participant.

Statistical analysis All analysis followed the Consolidated Standards of Reporting Trials (CONSORT) statement for randomized controlled trials. Statistical analyses were conducted following the intention-to-treat principle (ITT) using SPSS version 26. We used the multiple imputation (MI) procedure to impute missing sum scores for participants who did not complete the post- or six months follow-up assessments. MI is considered a to be a conservative approach for analysing incomplete datasets as it takes into account the uncertainty due to missing information. We used all available data from the pre-, post and six-months follow-up assessment as well as age, gender and educational level as predictors. Means, standard deviations, and standard errors of effect sizes were pooled from five sets of imputations. The effects of group on primary and secondary outcome measures of the ITT and completers-only datasets were analysed using repeated measures ANOVAs with time (pre, post and six-months follow-up) as a within-subject factor. Pooled F-values were calculated using RStudio. Cohen's d was reported for the between-group effect sizes and corresponding 95% confidence intervals (95% CI). Analysis of outcomes at baseline and demographical variables between complete and missing data were analysed using T- and Chi2-tests. Completers data on sickness absence and long-term sick leave were analysed using Kruskal-Wallis-test, non-parametric test recommended for comparison of three or more samples. To evaluate clinically significant change, we used the guidelines by Jacobson and Truax (1991). Clinically significant change was based on the completer's analysis. To meet the criteria for clinically significant change on the primary outcome SMBQ, participants had to demonstrate a reliable change of 0.69 and score under the cut-off of 4.4, in accordance with a recent study in a clinical sample by van de Leur et al. (2020). We completed the clinically significant change analysis with KEDS. On the KEDS, participants had to demonstrate a reliable change of 8.72 and score under the cut off of 19.

ELIGIBILITY:
Inclusion Criteria:

Participants were employees who had volunteered for the trial. To be eligible for the study, they had to fulfil the criteria for an adjustment disorder described in the subdivision F43 Reaction to severe stress, and adjustment disorders of the ICD-10. The diagnosis was established through telephone interviews using the Mini International Neuropsychiatric Interview, additional criteria from the International Statistical Classification of Diseases and Related Health Problems (ICD-10; 25), and national diagnostic guidelines regarding stress-related disorders.

In addition to an adjustment disorder, participants had to fulfil the following criteria: (i) a minimum age of 18 years, (ii) mastering Swedish, (iii) have access to a computer or a tablet computer with internet-access, (iv) currently employed, (v) score of >1.5 points on the Shirom Melamed Burnout Questionnaire (SMBQ), <34 points on the Montgomery Åsberg Depression Scale-Self Rated (MADRS-S), <21 points on the Insomnia Severity Index (ISI) and <14 points on the Alcohol Use Disorders Identification Test (AUDIT). Mild to moderate forms of DSM axis-I diagnosis were accepted as co-morbid conditions, as long as these were considered to be secondary to the primary adjustment disorder. Participants' on full- or part-time sick leave, one year or less, were also included.

Exclusion Criteria:

Participants were excluded from the study if they (i) currently in treatment for stress-related disorder, (ii) currently were suffering from bipolar disorder, psychosis, post-traumatic stress disorder (PTSD), eating disorder, substance abuse, severe forms of depression, anxiety disorder or personality disorders, or (iv) were showing suicidal ideation based on item 9 of the MADRS-S. Participants on medication (e.g., antidepressants or sleep medication) were not excluded from the study but were requested to keep their medication constant during the study period.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2017-01-20 (Actual); Primary Completion 2019-08-26 (Actual); Study Completion 2019-08-26 (Actual)

PRIMARY OUTCOMES:
Shirom-Melamed Burnout Questionnaire | Change between baseline and end of treatment after ten weeks and follow-up at 6 month and 1 year after treatment
  The Shirom-Melamed Burnout Questionnaire (SMBQ; Melamed et al., 1992, 1999), is a 22-item scale (graded 1-7) used to assess different aspects of chronic stress and burnout (Physical Fatigue, Cognitive weariness, Tension, and Listlessness). This scale correlates signiﬁcantly [58] with other well established questionnaires measuring burnout, e.g., Maslach Burnout Inventory [59]. The SMBQ has an internal consistency reliability (Cronbach's alpha) of .92. [56].

SECONDARY OUTCOMES:
Perceived Stress Scale | Change between baseline and end of treatment after ten weeks and follow-up at 6 month and 1 year after treatment
  Perceived stress was measured with the 10-item version of the Perceived Stress Scale (PSS-14), translated into Swedish [60,61]. The PSS-10 is designed to measure the degree to which situations in one's life are appraised as stressful. The Swedish version of PSS has an internal consistency reliability (Cronbach's alpha) of .82 and split-half reliability estimate of .84 [61].
Karolinska Exhaustion Disorder Scale | Change between baseline and end of treatment after ten weeks and follow-up at 6 month and 1 year after treatment
  Karolinska Exhaustion Disorder Scale (KEDS-9) is a 9-item questionnaire measuring symptoms of chronic stress, fatigue and exhaustion [62]. The instrument is answered on a 7-point scale, with a scale range of 0-54. A cut-off score of 19 was shown to discriminate between healthy subjects and patients with chronic stress and exhaustion [62]. KEDS-9 has satisfactory reliability, Cronbach's alpha of .94 [62].
Montgomery Åsberg Depression Rating Scale | Change between baseline and end of treatment after ten weeks and follow-up at 6 month and 1 year after treatment
  We used the Montgomery Åsberg Depression Rating Scale self-assessment, MADRS-S [63] to measure symptoms of depression. MADRS-S consists of nine items measuring different symptoms of depression and each symptom is rated on a six-point scale. The instrument has good reliability [64] and has been validated as an internet-based measure [65]. In a comparative study [66] the MADRS-S correlated highly (r = .87) with the Beck Depression Inventory [67], indicating acceptable convergent validity.
Generalised Anxiety Disorder Scale | Change between baseline and end of treatment after ten weeks and follow-up at 6 month and 1 year after treatment
  Generalized Anxiety Disorder 7-item Scale (GAD-7) is an instrument assessing excessive worry and generalized anxiety disorder. GAD-7 had good internal consistency reliability (α = .83), test-retest reliability (r = .83), as well as criterion, construct, factorial, and procedural validity [68]. A cut-off score of 10 has been suggested to discriminates between healthy subjects and patients with generalized anxiety disorder.
Insomnia Severity Index | Change between baseline and end of treatment after ten weeks and follow-up at 6 month and 1 year after treatment
  The Insomnia Severity Index (ISI) is a 7-item self-report questionnaire that measures individuals perceptions of their insomnia and the severity of problems with delayed sleep onset, sleep maintenance, and early morning awakenings [69]. ISI exhibits adequate internal consistency measures (α =.74), and is a sensitive measure to detect changes in perceived sleep difficulties [69]. It has previously been validated as an internet-based measure [70].
Alcohol Use Disorders Identification Test | Change between baseline and end of treatment after ten weeks
  The Alcohol Use Disorders Identification Test (AUDIT; [71] was used to assess potential alcohol dependence or abuse. In a study of the psychometric properties of the Swedish version of AUDIT, both internal and test-retest reliabilities were satisfactory [72]. A cut-off of <14 points on the AUDIT indicating risk of overconsumption of alcohol [73].
Work Experience Measurement Scale | Change between baseline and end of treatment after ten weeks and follow-up at 6 month and 1 year after treatment
  The Work Experience Measurement Scale (WEMS) is an instrument measuring the experience of work from a health resource perspective [74]. WEMS consists of 32 items measuring job satisfaction in five different domains (supportive work conditions, internal work experience, autonomy, time experience, management, process of change) on a six-point scale. Cronbach's alpha on the WEMS has been reported to be in the interval of .85-.96 [74].
Work Ability Index | Change between baseline and end of treatment after ten weeks and follow-up at 6 month and 1 year after treatment
  Work Ability Index (WAI) is an instrument for assessing health status and work ability among employees [75-77]. The WAI comprises of different scales, with scores ranging from 7 to 49 points. Studies [75] have suggested that 7-27 points = poor; 28-36 points = moderate; 37-43 points = good; and 44-49 points indicates excellent work ability. Analyses of reliability indicates satisfactory internal consistency, α-levels ranging from .79 to .80 [78,79].
Sheehan Disability Scale | Change between baseline and end of treatment after ten weeks and follow-up at 6 month and 1 year after treatment
  Sheehan Disability Scale (SDS) measures quality of life and everyday function in three domains; Work ability, Social life and Family life. The instrument is answered on a 10-point VAS scale, with a scale range of 0-30. SDS has satisfactory internal consistency reliability (α = 0.89) and test-retest reliability (r = 0.73; 42,43).
Recovery Experiences Questionnaire | Change between baseline and end of treatment after ten weeks and follow-up at 6 month and 1 year after treatment
  The 16-item Recovery Experience Questionnaire (REQ) includes four factors, representing four different recovery experiences; (i) psychological detachment (ii) relaxation, (iii) mastery and (iv) control [82]. The questionnaire is answered on a 5-point Likert scale, and has been validated in a Swedish population showing excellent internal consistency, α=0.92 [83].
Trimbos and Institute of Medical Technology Assessment Cost Questionnaire for Psychiatry | Change between baseline and end of treatment after ten weeks and follow-up at 6 month and 1 year after treatment
  TiC-P has been used in several studies for economic evaluations of healthcare consumption and productivity loss in mental health [84]. Sickness absence were conceptualized as the self-rated number of days during the past three months absent from work while being physically or mentally ill.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Behavioral Sciences and Learning, Linköping University, Linköping, Östergötland County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Eurofound. Sixth European Working Conditions Survey - Overview report (2017 update). Luxembourg: Publications Office of the European Union; 2017.
- [Background] World Health Organization. The global burden of disease : 2004 update. Geneva: World Health Organization; 2008.
- [Background] Sterling P, Eyer J. A new paradigm to explain arousal pathology. In: Fisher S, Reason J, editors. Handb Life Stress Cogn Health Oxford: John Wiley & Sons; 1988. p. xxxiii, 750.
- [Derived] Persson Asplund R, Asplund S, von Buxhoeveden H, Delby H, Eriksson K, Svenning Gerhardsson M, Palm J, Skyttberg T, Torstensson J, Ljotsson B, Carlbring P, Andersson G. Work-Focused Versus Generic Internet-Based Interventions for Employees With Stress-Related Disorders: Randomized Controlled Trial. J Med Internet Res. 2023 Apr 25;25:e34446. doi: 10.2196/34446. PMID 37097739